CLINICAL TRIAL: NCT01235793
Title: A Phase 2a Study of the Addition of Temozolomide to a Standard Conditioning Regimen for Autologous Stem Cell Transplantation in Relapsed and Refractory Central Nervous System (CNS) Lymphoma
Brief Title: The Addition of Temozolomide to Conditioning for Autologous Transplantation in Relapsed & Refractory CNS Lymphoma
Acronym: DRBEAT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The clinical trial was terminated due to poor enrollment
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Yuliya Linhares, Interim Lead Investigator, Staff Physician, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00019873
Record Dates: First submitted 2010-11-05; First posted 2010-11-08 (Estimated); Results first posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-10

CONDITIONS: B-Cell Lymphoma Originating in the CNS
Keywords: Relapsed; Refractory; Primary Central Nervous System B-cell Lymphoma; Autologous Stem Cell Transplant; Temozolomide; B-Cell Lymphoma; RBEAM; Conditioning Regimen
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DRBEAT Regimen (Experimental)
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide — The DRBEAT regimen will be similar to RBEAM. Rituximab and Carmustine will be given Day -6. Etoposide and Cytarabine will be given on Days -5 to -2. Temozolomide will be given via divided doses over five days starting on Day -5 to Day -1. A dose escalation design, known as EWOC (Escalation with overdose control) will be used to determine the target dose of temozolomide for this study. The starting dose given over five days will begin at 250mg/m2 (cumulative total dose of 1250 mg/m2), as previous data indicates this to be a safe dose. Based on the reported Dose Limiting toxicities from the previous patients, the EWOC statistical modeling will be performed to determine the next dose level.

SUMMARY:
The primary purpose of the study will be testing the dosing of temozolomide to find the target dose that a person can tolerate. The other part of the study will be determining how helpful it can be to CNS lymphoma patients by adding temozolomide to the "conditioning regimen" prior to stem cell transplantation.

This research study is designed to test the investigational use of temozolomide as part of a conditioning regimen prior to stem cell transplantation. This drug has not yet been approved by the U.S. Food and Drug Administration (FDA) to be used in the setting of stem cell transplantation in lymphomas of the brain (central nervous system or CNS) but it has been studied and used before in transplantation with reasonable results.

DETAILED DESCRIPTION:
Currently there is no standard of care for relapsed or refractory primary central nervous system (CNS) lymphoma. After high-dose methotrexate or radiation therapy, the best approach to relapsed disease is undefined. Common practice is the regimen RBEAM as a conditioning regimen in this patient population prior to transplantation. The RBEAM regimen includes R (rituximab), B (BCNU), E (etoposide), A (Ara-C (cytarabine)) and M (melphalan). In addition, dexamethasone is included in the regimen although not noted in the RBEAM mnemonic. However, the melphalan used in this combination is not thought to have much CNS penetration. Therefore, temozolomide, an alkylating agent known to penetrate the CNS and approved by the FDA for brain tumors will be used and evaluated in this study instead of melphalan.

The aim of this study is to determine an effective and safe dose of temozolomide orally administered to patients with relapsed primary CNS lymphoma over the 5 days preceding autologous stem-cell transplantation. The hope is that the conditioning regimen DRBEAT [D (dexamethasone) (R (rituximab), B (BCNU), E (etoposide), A (Ara-C (cytarabine)) and T (temozolomide)] will significantly improve the survival of patients with relapsed CNS lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age and ≤ 75 years of age
2. Patients must have Central Nervous System (CNS) involvement with a mature B-cell non-Hodgkin's Lymphoma, (WHO criteria)
3. Patients must meet one of the below criteria:

   * Patients who have achieved a complete response (CR) or partial response (PR) after initial therapy for Central Nervous System (CNS) B-cell lymphoma, OR
   * Patients with relapsed or progressed disease following therapy for CNS B-cell lymphoma who has achieved a subsequent CR or PR following salvage chemotherapy, OR
   * Patients who are initially refractory to therapy for CNS B-cell lymphoma but who have achieved a CR or PR following a salvage chemotherapy regimen, OR
   * Patients who have developed CNS relapse from systemic B-cell Non-Hodgkin's lymphoma, and have evidence of chemotherapy sensitive lymphoma.
4. Patients fit for autologous stem cell transplantation
5. Patients able to understand and willing to sign a written informed consent document

Exclusion Criteria:

1. Patients whose life expectancy is severely limited by diseases other than malignancy
2. Karnofsky Performance Score <60
3. Patients who are pregnant or breastfeeding
4. Patients who are HIV seropositive
5. Patients who have an uncontrolled infection (presumed or documented) with progression after appropriate therapy for greater than one month
6. Patients with symptomatic coronary artery disease, uncontrolled congestive heart failure. Left Ventricular Ejection Fraction is not required to be measured, however if it is measured, patient is excluded if ejection fraction is <30%
7. Patients requiring supplementary continuous oxygen. DLCO is not required to be measured, however if it is measured, patient is excluded if DLCO <35%.
8. Patients with clinical or laboratory evidence of liver disease will be evaluated for the cause of liver disease, its clinical severity in terms of liver function and histology, and for the degree of portal hypertension. Patients with any of the following liver function abnormalities will be excluded

   1. Fulminant liver failure
   2. Cirrhosis with evidence of portal hypertension or bridging fibrosis
   3. Alcoholic hepatitis
   4. Esophageal varices
   5. A history of bleeding esophageal varices
   6. Hepatic encephalopathy
   7. Uncorrectable hepatic synthetic dysfunction evidenced by prolongation of the prothrombin time
   8. Ascites related to portal hypertension
   9. Chronic viral hepatitis with total serum bilirubin >3 mg/dL
   10. Symptomatic biliary disease
9. Patients with non-B-cell lymphomas or brain tumors that are not lymphomas are Excluded from the study. Non-B-cell lymphomas include: any T-cell lymphoma, natural killer (NK)-cell lymphomas, and Hodgkin lymphomas
10. Patients for whom an insufficient number of stem cells (<2 X 106/kg) have been collected

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-10-14 (Actual); Primary Completion 2017-07-28 (Actual); Study Completion 2018-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lill, MD, Principal Investigator — Cedars-Sinai Medical Center; Yuliya Linhares, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Soussain C, Hoang-Xuan K, Taillandier L, Fourme E, Choquet S, Witz F, Casasnovas O, Dupriez B, Souleau B, Taksin AL, Gisselbrecht C, Jaccard A, Omuro A, Sanson M, Janvier M, Kolb B, Zini JM, Leblond V; Societe Francaise de Greffe de Moelle Osseuse-Therapie Cellulaire. Intensive chemotherapy followed by hematopoietic stem-cell rescue for refractory and recurrent primary CNS and intraocular lymphoma: Societe Francaise de Greffe de Moelle Osseuse-Therapie Cellulaire. J Clin Oncol. 2008 May 20;26(15):2512-8. doi: 10.1200/JCO.2007.13.5533. Epub 2008 Apr 14. PMID 18413641
- [Background] Sierra del Rio M, Rousseau A, Soussain C, Ricard D, Hoang-Xuan K. Primary CNS lymphoma in immunocompetent patients. Oncologist. 2009 May;14(5):526-39. doi: 10.1634/theoncologist.2008-0236. Epub 2009 May 11. PMID 19433528
- [Background] Soussain C, Suzan F, Hoang-Xuan K, Cassoux N, Levy V, Azar N, Belanger C, Achour E, Ribrag V, Gerber S, Delattre JY, Leblond V. Results of intensive chemotherapy followed by hematopoietic stem-cell rescue in 22 patients with refractory or recurrent primary CNS lymphoma or intraocular lymphoma. J Clin Oncol. 2001 Feb 1;19(3):742-9. doi: 10.1200/JCO.2001.19.3.742. PMID 11157026
- [Background] Cheng T, Forsyth P, Chaudhry A, Morris D, Gluck S, Russell JA, Stewart DA. High-dose thiotepa, busulfan, cyclophosphamide and ASCT without whole-brain radiotherapy for poor prognosis primary CNS lymphoma. Bone Marrow Transplant. 2003 Apr;31(8):679-85. doi: 10.1038/sj.bmt.1703917. PMID 12692608
- [Background] Abrey LE, Moskowitz CH, Mason WP, Crump M, Stewart D, Forsyth P, Paleologos N, Correa DD, Anderson ND, Caron D, Zelenetz A, Nimer SD, DeAngelis LM. Intensive methotrexate and cytarabine followed by high-dose chemotherapy with autologous stem-cell rescue in patients with newly diagnosed primary CNS lymphoma: an intent-to-treat analysis. J Clin Oncol. 2003 Nov 15;21(22):4151-6. doi: 10.1200/JCO.2003.05.024. PMID 14615443
- [Background] Colombat P, Lemevel A, Bertrand P, Delwail V, Rachieru P, Brion A, Berthou C, Bay JO, Delepine R, Desablens B, Camilleri-Broet S, Linassier C, Lamy T. High-dose chemotherapy with autologous stem cell transplantation as first-line therapy for primary CNS lymphoma in patients younger than 60 years: a multicenter phase II study of the GOELAMS group. Bone Marrow Transplant. 2006 Sep;38(6):417-20. doi: 10.1038/sj.bmt.1705452. PMID 16951691
- [Background] Mills W, Chopra R, McMillan A, Pearce R, Linch DC, Goldstone AH. BEAM chemotherapy and autologous bone marrow transplantation for patients with relapsed or refractory non-Hodgkin's lymphoma. J Clin Oncol. 1995 Mar;13(3):588-95. doi: 10.1200/JCO.1995.13.3.588. PMID 7884420
- [Background] Philip T, Guglielmi C, Hagenbeek A, Somers R, Van der Lelie H, Bron D, Sonneveld P, Gisselbrecht C, Cahn JY, Harousseau JL, et al. Autologous bone marrow transplantation as compared with salvage chemotherapy in relapses of chemotherapy-sensitive non-Hodgkin's lymphoma. N Engl J Med. 1995 Dec 7;333(23):1540-5. doi: 10.1056/NEJM199512073332305. PMID 7477169
- [Background] Nakasone H, Izutsu K, Wakita S, Yamaguchi H, Muramatsu-Kida M, Usuki K. Autologous stem cell transplantation with PCR-negative graft would be associated with a favorable outcome in core-binding factor acute myeloid leukemia. Biol Blood Marrow Transplant. 2008 Nov;14(11):1262-9. doi: 10.1016/j.bbmt.2008.08.012. PMID 18940681
- [Background] Gondo H, Harada M, Miyamoto T, Takenaka K, Tanimoto K, Mizuno S, Fujisaki T, Nagafuji K, Hayashi S, Eto T, Taniguchi S, Akashi K, Harada N, Yamasaki K, Shibuya T, Matsuishi E, Ohno Y, Makino S, Takamatsu Y, Murakawa M, Teshima T, Hirota Y, Okamura T, Kinukawa N, Niho Y, et al. Autologous peripheral blood stem cell transplantation for acute myelogenous leukemia. Bone Marrow Transplant. 1997 Nov;20(10):821-6. doi: 10.1038/sj.bmt.1700979. PMID 9404921
- [Background] Coiffier B, Lepage E, Briere J, Herbrecht R, Tilly H, Bouabdallah R, Morel P, Van Den Neste E, Salles G, Gaulard P, Reyes F, Lederlin P, Gisselbrecht C. CHOP chemotherapy plus rituximab compared with CHOP alone in elderly patients with diffuse large-B-cell lymphoma. N Engl J Med. 2002 Jan 24;346(4):235-42. doi: 10.1056/NEJMoa011795. PMID 11807147
- [Background] Jeffrey Raizer, DeAngelis Lisa, Andrew Zelenetz et al. Activity of Rituximab in Primary Central Nervous System Lymphoma PCNSL. Proc Am Soc Clin Oncol 19: 2000 (abstr 642)
- [Background] Rubenstein JL, Fridlyand J, Abrey L, Shen A, Karch J, Wang E, Issa S, Damon L, Prados M, McDermott M, O'Brien J, Haqq C, Shuman M. Phase I study of intraventricular administration of rituximab in patients with recurrent CNS and intraocular lymphoma. J Clin Oncol. 2007 Apr 10;25(11):1350-6. doi: 10.1200/JCO.2006.09.7311. Epub 2007 Feb 20. PMID 17312328
- [Background] Wong ET, Tishler R, Barron L, Wu JK. Immunochemotherapy with rituximab and temozolomide for central nervous system lymphomas. Cancer. 2004 Jul 1;101(1):139-45. doi: 10.1002/cncr.20339. PMID 15221999
- [Background] Enting RH, Demopoulos A, DeAngelis LM, Abrey LE. Salvage therapy for primary CNS lymphoma with a combination of rituximab and temozolomide. Neurology. 2004 Sep 14;63(5):901-3. doi: 10.1212/01.wnl.0000137050.43114.42. PMID 15365145
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Background] Stupp R, Hegi ME, Gilbert MR, Chakravarti A. Chemoradiotherapy in malignant glioma: standard of care and future directions. J Clin Oncol. 2007 Sep 10;25(26):4127-36. doi: 10.1200/JCO.2007.11.8554. PMID 17827463
- [Background] Batchelor T, Carson K, O'Neill A, Grossman SA, Alavi J, New P, Hochberg F, Priet R. Treatment of primary CNS lymphoma with methotrexate and deferred radiotherapy: a report of NABTT 96-07. J Clin Oncol. 2003 Mar 15;21(6):1044-9. doi: 10.1200/JCO.2003.03.036. PMID 12637469
- [Background] Agarwala SS, Kirkwood JM. Temozolomide, a novel alkylating agent with activity in the central nervous system, may improve the treatment of advanced metastatic melanoma. Oncologist. 2000;5(2):144-51. doi: 10.1634/theoncologist.5-2-144. PMID 10794805
- [Background] Agarwala SS, Reyderman L, Statkevich P et al Pharmacokinetic phase I study of temozolomide penetration into CSF in a patient with dural melanoma. Annals of Oncology, supplement 4 to volume 9, 1998, abstract 659 page 138
- [Background] Vassal G, Tranchand B, Valteau-Couanet D, Mahe C, Couanet D, Schoeppfer C, Grill J, Kalifa C, Hill C, Ardiet C, Hartmann O. Pharmacodynamics of tandem high-dose melphalan with peripheral blood stem cell transplantation in children with neuroblastoma and medulloblastoma. Bone Marrow Transplant. 2001 Mar;27(5):471-7. doi: 10.1038/sj.bmt.1702806. PMID 11313680
- [Background] Slevin ML, Piall EM, Aherne GW, Harvey VJ, Johnston A, Lister TA. Effect of dose and schedule on pharmacokinetics of high-dose cytosine arabinoside in plasma and cerebrospinal fluid. J Clin Oncol. 1983 Sep;1(9):546-51. doi: 10.1200/JCO.1983.1.9.546. PMID 6583325
- [Background] Capizzi RL, Yang JL, Cheng E, Bjornsson T, Sahasrabudhe D, Tan RS, Cheng YC. Alteration of the pharmacokinetics of high-dose ara-C by its metabolite, high ara-U in patients with acute leukemia. J Clin Oncol. 1983 Dec;1(12):763-71. doi: 10.1200/JCO.1983.1.12.763. PMID 6668493
- [Background] Relling MV, Mahmoud HH, Pui CH, Sandlund JT, Rivera GK, Ribeiro RC, Crist WM, Evans WE. Etoposide achieves potentially cytotoxic concentrations in CSF of children with acute lymphoblastic leukemia. J Clin Oncol. 1996 Feb;14(2):399-404. doi: 10.1200/JCO.1996.14.2.399. PMID 8636749
- [Background] Newton HB, Turowski RC, Stroup TJ, McCoy LK. Clinical presentation, diagnosis, and pharmacotherapy of patients with primary brain tumors. Ann Pharmacother. 1999 Jul-Aug;33(7-8):816-32. doi: 10.1345/aph.18353. PMID 10466912
- [Background] Skeel R. Antioneoplastic Drugs and Biologic Response Modifiers: Classification, Use, and Toxicity of Clinically Useful Agents. Pp64-66 in Handbook of Cancer Chemotherapy, 5th edition 1999, Editor Skeel R
- [Background] Brox LW, Gowans B, Belch A. L-phenylalanine mustard (melphalan) uptake and cross-linking in the RPMI 6410 human lymphoblastoid cell line. Cancer Res. 1980 Apr;40(4):1169-72. PMID 7357546
- [Background] Chabner B. Adduct-Forming Agents: Alkylating Agents and Platinum Analogs. Pp 52-53 in Harrison's Manual of Oncology 2008. Editors Chabner BA, Lynch TJ, Longo DL
- [Background] Gaspard MH, Maraninchi D, Stoppa AM, Gastaut JA, Michel G, Tubiana N, Blaise D, Novakovitch G, Rossi JF, Weiller PJ, et al. Intensive chemotherapy with high doses of BCNU, etoposide, cytosine arabinoside, and melphalan (BEAM) followed by autologous bone marrow transplantation: toxicity and antitumor activity in 26 patients with poor-risk malignancies. Cancer Chemother Pharmacol. 1988;22(3):256-62. doi: 10.1007/BF00273421. PMID 3044633
- [Background] Hoffmann AL, Buhk JH, Strik H. Neoplastic meningitis from breast cancer: feasibility and activity of long-term intrathecal liposomal Ara-C combined with dose-dense temozolomide. Anticancer Res. 2009 Dec;29(12):5191-5. PMID 20044635
- [Background] Passarin MG, Moretto G, Musso AM, Ottaviani S, Masotto B, Ghimenton C, Iuzzolino P, Buffone E, Ruda R, Soffietti R, Vattemi E, Pedersini R. Intrathecal liposomal cytarabine in combination with temozolomide in low-grade oligoastrocytoma with leptomeningeal dissemination. J Neurooncol. 2010 May;97(3):439-44. doi: 10.1007/s11060-009-0040-0. Epub 2009 Oct 31. PMID 19876600
- [Background] Issa S, Hwang J, Karch J, et al. Treatment of primary CNS lymphoma with induction high-dose methotrexate, temozolomide, rituximab followed by consolidation cytarabine/etoposide: A pilot study with biomarker analysis. Journal of Clinical Oncology, 2006 ASCO Annual Meeting Proceedings Part I. Vol 24, No. 18S (June 20 Supplement), 2006: 7595
- [Background] Prados MD, Yung WK, Fine HA, Greenberg HS, Junck L, Chang SM, Nicholas MK, Robins HI, Mehta MP, Fink KL, Jaeckle KA, Kuhn J, Hess KR, Schold SC Jr; North American Brain Tumor Consortium study. Phase 2 study of BCNU and temozolomide for recurrent glioblastoma multiforme: North American Brain Tumor Consortium study. Neuro Oncol. 2004 Jan;6(1):33-7. doi: 10.1215/S1152851703000309. PMID 14769138
- [Background] Raizer JJ, Malkin MG, Kleber M, Abrey LE. Phase 1 study of 28-day, low-dose temozolomide and BCNU in the treatment of malignant gliomas after radiation therapy. Neuro Oncol. 2004 Jul;6(3):247-52. doi: 10.1215/S1152851704000122. PMID 15279717
- [Background] Ebert BL, Niemierko E, Shaffer K, Salgia R. Use of temozolomide with other cytotoxic chemotherapy in the treatment of patients with recurrent brain metastases from lung cancer. Oncologist. 2003;8(1):69-75. doi: 10.1634/theoncologist.8-1-69. PMID 12604733
- [Background] Korones DN, Benita-Weiss M, Coyle TE, Mechtler L, Bushunow P, Evans B, Reardon DA, Quinn JA, Friedman H. Phase I study of temozolomide and escalating doses of oral etoposide for adults with recurrent malignant glioma. Cancer. 2003 Apr 15;97(8):1963-8. doi: 10.1002/cncr.11260. PMID 12673724
- [Background] Rudek MA, Donehower RC, Statkevich P, Batra VK, Cutler DL, Baker SD. Temozolomide in patients with advanced cancer: phase I and pharmacokinetic study. Pharmacotherapy. 2004 Jan;24(1):16-25. doi: 10.1592/phco.24.1.16.34800. PMID 14740784
- [Background] Vera K, Djafari L, Faivre S, Guillamo JS, Djazouli K, Osorio M, Parker F, Cioloca C, Abdulkarim B, Armand JP, Raymond E. Dose-dense regimen of temozolomide given every other week in patients with primary central nervous system tumors. Ann Oncol. 2004 Jan;15(1):161-71. doi: 10.1093/annonc/mdh003. PMID 14679137
- [Background] Dhodapkar M, Rubin J, Reid JM, Burch PA, Pitot HC, Buckner JC, Ames MM, Suman VJ. Phase I trial of temozolomide (NSC 362856) in patients with advanced cancer. Clin Cancer Res. 1997 Jul;3(7):1093-100. PMID 9815788
- [Background] Handbook of statistics in clinical oncology By John Crowley, Donna Pauler Ankerst Pahse 1 Trials Page 8 Edition 2, 2005
- [Background] Hahn T, Wolff SN, Czuczman M, Fisher RI, Lazarus HM, Vose J, Warren L, Watt R, McCarthy PL Jr; ASBMT Expert Panel. The role of cytotoxic therapy with hematopoietic stem cell transplantation in the therapy of diffuse large cell B-cell non-Hodgkin's lymphoma: an evidence-based review. Biol Blood Marrow Transplant. 2001;7(6):308-31. doi: 10.1016/s1083-8791(01)80003-3. No abstract available. PMID 11464975
- [Background] Abrey LE, Batchelor TT, Ferreri AJ, Gospodarowicz M, Pulczynski EJ, Zucca E, Smith JR, Korfel A, Soussain C, DeAngelis LM, Neuwelt EA, O'Neill BP, Thiel E, Shenkier T, Graus F, van den Bent M, Seymour JF, Poortmans P, Armitage JO, Cavalli F; International Primary CNS Lymphoma Collaborative Group. Report of an international workshop to standardize baseline evaluation and response criteria for primary CNS lymphoma. J Clin Oncol. 2005 Aug 1;23(22):5034-43. doi: 10.1200/JCO.2005.13.524. Epub 2005 Jun 13. PMID 15955902
- [Background] Patel M, McCully C, Godwin K, Balis FM. Plasma and cerebrospinal fluid pharmacokinetics of intravenous temozolomide in non-human primates. J Neurooncol. 2003 Feb;61(3):203-7. doi: 10.1023/a:1022592913323. PMID 12675312
- [Background] Ostermann S, Csajka C, Buclin T, Leyvraz S, Lejeune F, Decosterd LA, Stupp R. Plasma and cerebrospinal fluid population pharmacokinetics of temozolomide in malignant glioma patients. Clin Cancer Res. 2004 Jun 1;10(11):3728-36. doi: 10.1158/1078-0432.CCR-03-0807. PMID 15173079
- [Background] Lowsky et al. Research Protocol for California AML Study.
- [Background] Babb J, Rogatko A, Zacks S. Cancer phase I clinical trials: efficient dose escalation with overdose control. Stat Med. 1998 May 30;17(10):1103-20. doi: 10.1002/(sici)1097-0258(19980530)17:103.0.co;2-9. PMID 9618772
- [Background] Babb JS, Rogatko A. Patient specific dosing in a cancer phase I clinical trial. Stat Med. 2001 Jul 30;20(14):2079-90. doi: 10.1002/sim.848. PMID 11439422
- [Background] Tighiouart M, Rogatko A, Babb JS. Flexible Bayesian methods for cancer phase I clinical trials. Dose escalation with overdose control. Stat Med. 2005 Jul 30;24(14):2183-96. doi: 10.1002/sim.2106. PMID 15909291
- [Background] Zacks s, Rogatko A, Babb J. Optimal Bayesian-feasible dose escalation for cancer phase I trials. Statistics & Probability Letters, 1998, vol. 38, issue 3, pages 215-220
- [Background] Xu Z, Tighiouart M, Rogatko A. 2007 EWOC 2.0: Interactive Software for Dose Escalation in Cancer Phase I Clinical Trials, Drug Information Journal, 41(2):221-228
- [Background] Chao ST, Barnett GH, Vogelbaum MA, Angelov L, Weil RJ, Neyman G, Reuther AM, Suh JH. Salvage stereotactic radiosurgery effectively treats recurrences from whole-brain radiation therapy. Cancer. 2008 Oct 15;113(8):2198-204. doi: 10.1002/cncr.23821. PMID 18780319
- [Background] Boiardi A, Silvani A, Pozzi A, Salmaggi A. Radiotherapy at tumor recurrence in primary CNS lymphoma. Neurology. 1998 Jun;50(6):1934-5. doi: 10.1212/wnl.50.6.1934-b. No abstract available. PMID 9633783
- [Background] Plotkin SR, Betensky RA, Hochberg FH, Grossman SA, Lesser GJ, Nabors LB, Chon B, Batchelor TT. Treatment of relapsed central nervous system lymphoma with high-dose methotrexate. Clin Cancer Res. 2004 Sep 1;10(17):5643-6. doi: 10.1158/1078-0432.CCR-04-0159. PMID 15355887
- [Background] Voloschin AD, Betensky R, Wen PY, Hochberg F, Batchelor T. Topotecan as salvage therapy for relapsed or refractory primary central nervous system lymphoma. J Neurooncol. 2008 Jan;86(2):211-5. doi: 10.1007/s11060-007-9464-6. Epub 2007 Sep 21. PMID 17896078
- [Background] Reni M, Mazza E, Foppoli M, Ferreri AJ. Primary central nervous system lymphomas: salvage treatment after failure to high-dose methotrexate. Cancer Lett. 2007 Dec 18;258(2):165-70. doi: 10.1016/j.canlet.2007.10.009. Epub 2007 Nov 13. PMID 17993246
- [Background] Reni M, Zaja F, Mason W, Perry J, Mazza E, Spina M, Bordonaro R, Ilariucci F, Faedi M, Corazzelli G, Manno P, Franceschi E, Pace A, Candela M, Abbadessa A, Stelitano C, Latte G, Ferreri AJ. Temozolomide as salvage treatment in primary brain lymphomas. Br J Cancer. 2007 Mar 26;96(6):864-7. doi: 10.1038/sj.bjc.6603660. Epub 2007 Feb 27. PMID 17325700
- See also: Related Info — http://www.pfizer.ca
- See also: Related Info — http://www.accessdata.fda.gov/drugsatfda_docs/label/2003/20207slr007_alkeran_lbl.pdf
- See also: Related Info — http://www.uptodate.com
- See also: CTCAE version 4.03 — https://evs.nci.nih.gov/ftp1/CTCAE/CTCAE_4.03/CTCAE_4.03_2010-06-14_QuickReference_5x7.pdf
- See also: Related Info — http://www.uptodate.com/online/content/topic.do?topicKey=drug_a_k/74688&selectedTitle=1%7E150&source=search_result
- See also: Related Info — http://www.accessdata.fda.gov/drugsatfda_docs/label/2009/103705s5299lbl.pdf
- See also: Related Info — http://www.accessdata.fda.gov/drugsatfda_docs/label/2007/017422s037lbl.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- DRBEAT Regimen: Temozolomide: The DRBEAT regimen will be similar to RBEAM. Rituximab and Carmustine will be given Day -6. Etoposide and Cytarabine will be given on Days -5 to -2. Temozolomide will be given via divided doses over five days starting on Day -5 to Day -1. A dose escalation design, known as EWOC (Escalation with overdose control) will be used to determine the target dose of temozolomide for this study. The starting dose given over five days will begin at 250mg/m^2 (cumulative total dose of 1250 mg/m^2), as previous data indicates this to be a safe dose. Based on the reported Dose Limiting toxicities from the previous patients, the EWOC statistical modeling will be performed to determine the next dose level.
Period: Overall Study
Arm/Group | DRBEAT Regimen
Started | 11
Completed | 5
Not Completed | 6
Not completed — Death | 6

BASELINE CHARACTERISTICS:
Arm/Group | DRBEAT Regimen
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 6
Age, Continuous [Median (Full Range); unit: Age in years] | 58 [32 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: One-year Progression-free Survival and Overall Survival
Description: Efficacy of the DRBEAT Regimen will be assessed by analysis of
  1. one-year progression-free survival (PFS), defined as the time interval from maximal response from therapy to tumor regrowth, progression*, or death, (*Progression is defined as meeting the response criteria listed in Table 4: Response Criteria for Primary Central Nervous System Lymphoma according to Abrey LE, Batchelor TT, Ferreri AJM et al.)
     and
  2. Overall survival, defined as the time interval between the date of transplant and the date of death from any cause.
Time Frame: (1) One Year (2) Until date of death from any cause, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | DRBEAT Regimen
Number analyzed (Participants) | 11
Days
  Progression Free Survival | 132 [38 to NA] — 95% confidence interval upper bound not obtained (insufficient number of participants with events)
  Overall Survival | 564 [71 to NA] — 95% confidence interval upper bound not obtained (insufficient number of participants with events)

2. Primary Outcome: Safest Dose of Temozolomide for the DRBEAT Regimen
Description: Safety will be assessed using a dose escalation design for temozolomide's use to determine the target dose and also to evaluate any and all acute treatment related toxicities. During the course of patient follow up and therapy, toxicities will be evaluated, particularly as the investigators will be determining the target dose of temozolomide. One of the major criteria for dose limiting toxicity for the study will be any Grade 3 or 4 nonhematologic toxicity from a list of commonly expected toxicities associated with autologous transplantation and temozolomide.
Time Frame: One Year
Measure: Number (95% Confidence Interval); unit: dose in mg/m^2
Arm/Group | DRBEAT Regimen
Number analyzed (Participants) | 11
dose in mg/m^2 | 773.25 [496.38 to 1000]

ADVERSE EVENTS:
Time Frame: Over a two year period, from start of research therapy to 2 years post treatment.
Arm/Group | DRBEAT Regimen
All-Cause Mortality (participants affected / at risk) | 6/11
Serious Adverse Events (participants affected / at risk) | 6/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DRBEAT Regimen (N=11)
Encephalopathy (Nervous system disorders) | 1 (1) — Temozolomide 431 mg/m^2
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) — Temozolomide 351 mg/m^2
Gait disturbances (Nervous system disorders) | 1 (1) — Temozolomide 431 mg/m^2
Renal and Urinary disorders -Other, specify: High squamous epithelial cells (Renal and urinary disorders) | 1 (1) — Temozolomide 250 mg/m^2
Sepsis (Infections and infestations) | 3 (3) — Temozolomide 379 mg/m^2, 611 mg/m^2, and 762 mg/m^2
OTHER ADVERSE EVENTS (reported when occurring in more than 05% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DRBEAT Regimen (N=11)
Alanine aminotransferase increased (Investigations) | 1 (1) — Temozolomide 351 mg/m^2
Alkaline phosphatase increased (Investigations) | 1 (1) — Temozolomide 351 mg/m^2
Allergic reaction (Immune system disorders) | 1 (1) — Temozolomide 734 mg/m^2
Anemia (Blood and lymphatic system disorders) | 5 (5) — Temozolomide 379 mg/m^2, 521 mg/m^2, 611 mg/m^2, 734 mg/m^2, and 762 mg/m^2
Aspartate aminotransferase increased (Investigations) | 1 (1) — Temozolomide 351 mg/m^2
Blood and lymphatic disorders -Other, specify: Pancytopenia (Blood and lymphatic system disorders) | 1 (1) — Temozolomide 440 mg/m^2
Blood bilirubin increased (Investigations) | 2 (2) — Temozolomide 351 mg/m^2
Facial muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) — Temozolomide 379 mg/m^2
Fatigue (General disorders) | 2 (2) — Temozolomide 250 mg/m^2 and 431 mg/m^2
Febrile neutropenia (Blood and lymphatic system disorders) | 9 (11) — Temozolomide 250 mg/m^2 -1 participant, 287 mg/m^2 -1 participant, 351 mg/m^2 -1 participant (2 events), 379 mg/m^2 -1 participant (2 events), 431 mg/m^2 -1 participant, 521 mg/m^2 -1 participant, 611 mg/m^2 -1 participant, 693 mg/m^2 -1 participant
Hypertryglyceridemia (Metabolism and nutrition disorders) | 1 (1) — Temozolomide 734 mg/m^2
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) — Temozolomide 440 mg/m^2
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) — Temozolomide 250 mg/m^2 and 287 mg/m^2
Hypotension (Vascular disorders) | 1 (1) — Temozolomide 762 mg/m^2
Infections and infestations -Other, specify: Ecoli bacteria (Infections and infestations) | 1 (1) — Temozolomide 250 mg/m^2
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) — Temozolomide 521 mg/m^2
Lung infection (Infections and infestations) | 1 (1) — Temozolomide 762 mg/m^2
Lymphocyte count decreased (Investigations) | 3 (5) — Temozolomide 250 mg/m^2 -1 participant, 287 mg/m^2 -1 participant (2 events), and 431 mg/m^2 -1 participant (2 events)
Mucositis oral (Gastrointestinal disorders) | 1 (1) — Temozolomide 762 mg/m^2
Musculoskeletal and connective tissue disorders -Other, specify: Neck weakness (Musculoskeletal and connective tissue disorders) | 1 (1) — Temozolomide 379 mg/m^2
Neutrophil count decreased (Investigations) | 3 (5) — Temozolomide 250 mg/m^2 -1 participant, 351 mg/m^2 -1 participant (2 events), and 693 mg/m^2 -1 participant
Platelet count decreased (Investigations) | 9 (10) — Temozolomide 250 mg/m^2 -1 participant, 287 mg/m^2 -1 participant, 351 mg/m^2 -1 participant, 379 mg/m^2 -1 participant, 431 mg/m^2 -1 participant, 521 mg/m^2 -1 participant, 611 mg/m^2 -1 participant, 693 mg/m^2, 734 mg/m^2 -1 participant (2 events)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) — Temozolomide 693 mg/m^2
Somnolence (Nervous system disorders) | 1 (1) — Temozolomide 379 mg/m^2
Urinary incontinence (Renal and urinary disorders) | 1 (1) — Temozolomide 431 mg/m^2
Urinary tract infection (Renal and urinary disorders) | 3 (5) — Temozolomide 287 mg/m^2 -1 participant, 351 mg/m^2 -1 participant (3 events), and 611 mg/m^2 -1 participant
White blood cell decreased (Investigations) | 5 (9) — Temozolomide 250 mg/m^2 -1 participant, 287 mg/m^2 -1 participant, 351 mg/m^2 -1 participant (4 events), 431 mg/m^2 -1 participant, and 762 mg/m^2 -1 participant (2 events)

LIMITATIONS AND CAVEATS:
Enrollment in the clinical trial did not reach the target number of subjects needed to achieve target power and is insufficient to produce statistically reliable results. Clinical trial terminated due to poor enrollment but the outcomes are measured.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-19): https://cdn.clinicaltrials.gov/large-docs/93/NCT01235793/Prot_SAP_000.pdf